CLINICAL TRIAL: NCT04565873
Title: Thyroid Stimulating Hormone (TSH) Level Variations in Early Pregnancy and Feto-maternal Outcome; Retrospective Study.
Brief Title: Thyroid Stimulating Hormone (TSH) Level Variations in Early Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Naser Al-Husban, Assistant Professor, University of Jordan
Other Study IDs: retrospective study
Record Dates: First submitted 2020-09-09; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy Early; Pregnancy Related; Thyroid Dysfunction
Keywords: TSH; pregnancy; Fetal outcome; maternal outcome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- P1: Primigravida in group 1
  Interventions: Diagnostic Test: TSH
- M1: Multipara in group 1
  Interventions: Diagnostic Test: TSH
- P2: Primigravida in group 2
  Interventions: Diagnostic Test: TSH
- M2: Multipara in group 2
  Interventions: Diagnostic Test: TSH

INTERVENTIONS:
Diagnostic Test: TSH — retrospective TSH level

SUMMARY:
Retrospective comparative study comparing group 1 (TSH level 0.1-1.99 mIU/L) and group 2 (TSH level 2.0-4 mIU/L). Each group was further subdivided into primigravidae and multipara. 1527 pregnant women were included.

DETAILED DESCRIPTION:
This was a retrospective comparative study spanning January 2014 to December 2018. It was conducted at Jordan university hospital, a teaching referral hospital affiliated to the University of Jordan, Amman, Jordan. Pregnant patients, both primigravida and multipara who had a spontaneous singleton pregnancy with documented TSH level in the first 16 weeks' gestation were included. The investigators excluded all patients who had known thyroid dysfunction whether on treatment or not, molar pregnancies, multiple pregnancies, patients with hyperemesis gravidarum, all patients with anti-thyroid antibodies (Anti-TPO), patients with TSH ˃ 4.0 mIU/L or ˂ 0.1 mIU/L. This range was used as TSH ˂ 0.1 mIU/L indicated an undiagnosed subclinical hyperthyroidism and TSH ˃4.0 indicated undiagnosed hypothyroidism. In addition, there were wide variations in the TSH reference ranges. Participants' data were collected retrospectively from antenatal clinic notes, admission notes, labor ward and operative notes. Data included patients ID number, age, parity, body mass index (BMI) in kg/m2, TSH values in the first 16 weeks of pregnancy. The participants were divided into 2 groups according to their TSH values. Group one with TSH values between 0.1-1.99 mIU/L. Group 2 had TSH values between 2-4 mIU/L. Each group was then subdivided into 2 subgroups; primigravida and multipara. Group P1: Primigravida in group 1, Group P2: Primigravida in group 2, Group M1: Multiparous in group 1, Group M2: Multiparous in group 2.

The investigators calculated the mean, median and range of TSH in each subgroup. The feto-maternal outcome was then compared between the 2 groups. The investigators studied miscarriage rate, ectopic pregnancy rate, maternal blood sugar values (Fasting blood sugar (FBS), glucose tolerance test (GTT), HbA1c or a combination) between 26 and 34 weeks, development of high blood pressure at delivery, duration of pregnancy (gestational age at delivery), preterm delivery rate, abruption placenta, mode of delivery, birth weight and APGAR score at 1 and 5 minutes. Gestational diabetes mellitus (GDM) was diagnosed as an FBS 92-125 mg/dL or 1-hour plasma glucose levels of 180 or more following 75-gram oral glucose load or 2-hour plasma glucose 153-199 mg/dL. The study obtained the approval of the institutional review board (IRB) at Jordan University Hospital (JUH) number 179/2019 dated 17/4/2019.

The statistical analysis was performed with the Data Toolkit in Excel (Microsoft, Redmond, WA, USA) using descriptive analysis. Relative risk and 95% confidence intervals were also calculated to compare variables. P values were considered significant at ˂0.05. The obtained data were examined using a frequency table and are presented as frequency, percentage and mean

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women
2. Previously healthy

Exclusion Criteria:

1. known thyroid diseases

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant patients
Study Population: pregnant unknown to have thyroid disease
Sampling Method: Non-Probability Sample
Enrollment: 1527 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Feto-maternal outcome | 4 years
  miscarriage rate, preterm delivery,

CONTACTS AND LOCATIONS:
Overall Officials: Al-Husban Naser, Principal Investigator — The University of Jordan
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
retrospective; data are available on reasonable request